CLINICAL TRIAL: NCT05500456
Title: Evaluation of the Achieved Occlusal Relationships Using the PAR Index Between the In-house Constructed Clear Aligners and Fixed Appliances in Patients With Extraction-based Treatment Plans: A Randomized Control Clinical Trial
Brief Title: The Effectiveness of Clear Aligner and Traditional Fixed Appliances in Achieving Good Occlusion in Complex Orthodontic Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-13-2022
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Crowding, Tooth
Keywords: Clear aligners; PAR index; Vestibular fixed appliances; Orthodontics; Crowding; Treatment duration
MeSH Terms: conditions — Malocclusion; Crowding | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clear aligners (Experimental): The patients in this group will be treated using clear aligners.
  Interventions: Device: Clear aligners
- Fixed appliances. (Active Comparator): The patients in this group will be treated using fixed appliances.
  Interventions: Device: Fixed appliances

INTERVENTIONS:
Device: Clear aligners — Each aligner will be worn for about two weeks, and then replaced by the next in the series until the final position is achieved.
  Arms: Clear aligners
Device: Fixed appliances — Conventional wires and brackets will be used.
  Arms: Fixed appliances.

SUMMARY:
Patients who have severe crowding that requires four premolars extraction will be treated in this study. The efficacy and effectiveness of in-house clear aligners therapy compared with vestibular fixed appliances in the treatment of severe crowding malocclusion cases requiring the extraction of first premolars will be evaluated using Little's irregularity index (LII), Peer assessment rating index (PAR), and treatment duration.

There are two groups:

First group (Experimental): the patients in this group will be treated using clear aligners.

Second group (Control): the patients in this group will be treated using fixed appliances.

DETAILED DESCRIPTION:
For years, orthodontists and dentists have used removable appliances for orthodontic treatment. With the CAD/CAM technology, clear aligners treat a broader range of cases with greater precision. They consist of a series of plastic aligners that are intended to replace conventional wire and bracket technology for many orthodontic cases. Each custom-manufactured aligner exerts gentle, continuous forces to move teeth incrementally from their original state to a final, treated state. Each aligner is worn for about two weeks, then replaced by the next in the series until the final position is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Class I skeletal and dental malocclusion
* severe crowding (more than 6 mm of tooth size-arch length discrepancy)
* Good oral hygiene and periodontal health.
* No congenitally missing or extracted teeth (except for the third molars).
* No history of previous trauma to the maxillofacial region or surgical interventions.

Exclusion Criteria:

* Subject with psychological abnormalities.
* Subject with systemic diseases.
* Previous orthodontic treatment.
* Subject has known allergy to latex and plastic

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-05-11 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Change in PAR index | T0: one day before the commencement of treatment. T1: one day following the end of treatment
  The PAR index will be used to provide objective assessment of treatment success. Each set of dental models prepared before and after treatment for each case will be occluded in maximum intercuspation and a calibrated PAR ruler is used to assign a value to each of the PAR index components: contact displacement in the upper and lower labial segment (UAS), overjet (OJ), overbite (OB), medline deviation (MID) and right and left buccazzzl occlusion (RBO, LBO). The score of each component is summed up to a total PAR score. A reduction in the PAR score of at least 30% classifies the case as 'improved'. A reduction of 22 points or more in the weighted PAR score classifies the case as 'greatly improved'. Improvements smaller than 30% are declared as 'worse or no different'
Changes in Little's irregularity index | T0: one day before the commencement of treatment. T1: one day following the end of treatment
  The Little's index measures the linear displacements in the horizontal plane between the contact points of the anterior teeth from the mesial surface of one canine to the contralateral one. The LII score is the sum of these linear measurements, and a higher score value indicates more severe irregularities of the anterior teeth

SECONDARY OUTCOMES:
Treatment time | T1: one day following the end of treatment
  The treatment duration was calculated by months and will be compared between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Samer T Jaber, DDS,MSc, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y Hajeer, DDS,MSc,PhD, Study Director — Professor of Orthodontics, Department of Orthodontics, University of Damascus Dental School, Damascus, Syria.
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaber ST, Hajeer MY, Burhan AS, Latifeh Y. The Effect of Treatment With Clear Aligners Versus Fixed Appliances on Oral Health-Related Quality of Life in Patients With Severe Crowding: A One-Year Follow-Up Randomized Controlled Clinical Trial. Cureus. 2022 May 30;14(5):e25472. doi: 10.7759/cureus.25472. eCollection 2022 May. PMID 35663697
- [Background] Jaber ST, Hajeer MY, Khattab TZ, Mahaini L. Evaluation of the fused deposition modeling and the digital light processing techniques in terms of dimensional accuracy of printing dental models used for the fabrication of clear aligners. Clin Exp Dent Res. 2021 Aug;7(4):591-600. doi: 10.1002/cre2.366. Epub 2020 Nov 30. PMID 33258297
- [Background] Li W, Wang S, Zhang Y. The effectiveness of the Invisalign appliance in extraction cases using the the ABO model grading system: a multicenter randomized controlled trial. Int J Clin Exp Med. 2015 May 15;8(5):8276-82. eCollection 2015. PMID 26221410
- [Background] Liu S, Oh H, Chambers DW, Baumrind S, Xu T. Validity of the American Board of Orthodontics Discrepancy Index and the Peer Assessment Rating Index for comprehensive evaluation of malocclusion severity. Orthod Craniofac Res. 2017 Aug;20(3):140-145. doi: 10.1111/ocr.12195. Epub 2017 Jul 3. PMID 28670875
- [Background] KESLING HD. Coordinating the predetermined pattern and tooth positioner with conventional treatment. Am J Orthod Oral Surg. 1946 May;32:285-93. doi: 10.1016/0096-6347(46)90053-1. No abstract available. PMID 21027613